CLINICAL TRIAL: NCT01703819
Title: Efficacy Profile of Neurexan® in an Experimental Acute Stress Setting - an Explorative Double-blind Study in Healthy Probands
Brief Title: Explorative Efficacy Profile of Neurexan® in an Experimental Acute Stress Setting in Healthy Subjects
Acronym: NEUPRO-DB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1201; 2012-002358-22 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Acute Stress Reaction
Keywords: acute stress reaction; stress; stress perception; physiological stress response; Neurexan
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute | interventions — neurexan; stearic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurexan® (Experimental): 0.6 mg / tablet, 6 tablets, 1 tablet every 30 minutes from -180 minutes to -30 minutes
  Interventions: Drug: Neurexan®
- Placebo (Placebo Comparator): 6 tablets, 1 tablet every 30 minutes from -180 minutes to -30 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Neurexan® — 0.6 mg / tablet, 6 tablets, 1 tablet every 30 minutes from -180 minutes to -30 minutes
  Arms: Neurexan®
Other: Placebo — 6 tablets, 1 tablet every 30 minutes from -180 minutes to -30 minutes
  Other Names: Lactose monohydrate, magnesium stearate.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of acutely dosed Neurexan using an experimental stress test called the Trier Social Stress Test

DETAILED DESCRIPTION:
An acute stress reaction is a biopsychological condition arising in response to an event which is individually regarded as emotionally stressful. The onset of a stress response is associated with specific physiological actions in the sympathetic nervous system, both directly and indirectly through the release of adrenaline and to a lesser extent noradrenaline from the medulla of the adrenal glands. These catecholamine hormones facilitate immediate physical reactions by triggering increases in heart rate and breathing, constricting blood vessels. The other major player in the acute stress response is the hypothalamic-pituitary-adrenal axis.

Although stress has been described as a non-specific psychophysiological response to environmental stimuli, it is possible to discern specific bodily stress responses caused by specific emotional reactions to novel, ambivalent or uncontrollable situations and stimuli. For example, social stress induces elevated cortisol levels, particularly if the stressor is uncontrollable, unpredictable, and constitutes a social-evaluative threat due to the judgment of others such as in the Trier Social Stress Test. Usually, the TSST induces a two-fold increase in saliva cortisol with peaks around 10-20 min. after stress test termination. Also, an average increase in heart rates of around 20 beats per minute (bpm) is observed during the TSST. In addition, emotional states and feelings have been shown to be affected by this stress test, such as marked increases in stress perception,anxiety and emotional insecurity as well as decreases in mood, calmness and feeling awake.

Preliminary results indicate that Neurexan® may improve coping abilities in stressful situations. This study aims to investigate the effect of Neurexan® on subjectively perceived nervousness and tension during an acute stressful situation and to characterize the efficacy profile of Neurexan®.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Healthy male or female
3. age between 31 to 59 years
4. Fluent in German language.
5. Ability to understand the explanations and instructions given by the study physician

Exclusion Criteria:

1. allergies to ingredients of Neurexan® (Passiflora incarnata, Avena sativa, Coffea arabica, Zincum isovalerianicum, lactose monohydrate, magnesium stearate) or Placebo
2. lactose intolerance
3. use of any psychological stress-management intervention within the last 4 weeks
4. sick leave for any reason
5. participation in any other clinical study 3 months prior to Screening Visit
6. current or recent (3 months prior to Screening Visit) history of substance abuse or drug dependence including nicotine and alcohol (as verified in the respective IDCL list)
7. smokers
8. alcohol intake within last 24 hours (before Baseline Visit V3)
9. shift workers or work regularly during night time
10. use of any psychotropic medication or suffering from severe psychiatric illness needing acute intervention
11. BMI > 30 kg/m2
12. currently pregnant (verified by urine pregnancy test) or lactating
13. participation in a previous TSST study
14. high chronic stress as verified with the TICS-SSCS (a score of ≥ 23 on the screening scale for chronic stress meets the criterion of being chronically stressed)
15. major mental disorder as verified with the IDCL (depressive episode, panic disorder, social phobia, obsessive-compulsory disorder; alcohol dependency; schizophrenia and mania.)
16. employee of the Sponsor, one of the investigators or the CRO
17. use of any concomitant medication except contraceptives
18. any somatic disease or other condition the Investigator or their duly assigned representatives believes may affect the ability of the individual to complete the study or the interpretation of the study results
19. Individuals whose ability to speak for themselves lacks or can be doubted

Ages: 31 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Schedlowski, PhD, Principal Investigator — Institut für Medizinische Psychologie und Verhaltensimmunbiologie Universitätsklinikum Essen
Locations (2):
- Germany (2):
  - Institut fur Medizinische Psychologie und Verhaltensimmunbiologie Universitatsklinikum Essen, Essen
  - Klinische Psychologie und Psychotherapie, Fachbereich Psychologie, Universität Marburg, Marburg

REFERENCES:
- [Background] McEwen BS. Physiology and neurobiology of stress and adaptation: central role of the brain. Physiol Rev. 2007 Jul;87(3):873-904. doi: 10.1152/physrev.00041.2006. PMID 17615391
- [Background] Elsenbruch S, Lucas A, Holtmann G, Haag S, Gerken G, Riemenschneider N, Langhorst J, Kavelaars A, Heijnen CJ, Schedlowski M. Public speaking stress-induced neuroendocrine responses and circulating immune cell redistribution in irritable bowel syndrome. Am J Gastroenterol. 2006 Oct;101(10):2300-7. doi: 10.1111/j.1572-0241.2006.00837.x. Epub 2006 Sep 4. PMID 16952284
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Hellhammer J, Schubert M. The physiological response to Trier Social Stress Test relates to subjective measures of stress during but not before or after the test. Psychoneuroendocrinology. 2012 Jan;37(1):119-24. doi: 10.1016/j.psyneuen.2011.05.012. PMID 21689890
- [Background] Schult J, Hero T, Hellhammer J. Effects of powdered fertilized eggs on the stress response. Clin Nutr. 2010 Apr;29(2):255-60. doi: 10.1016/j.clnu.2009.09.004. Epub 2009 Oct 17. PMID 19837490
- [Background] Mason JW. A review of psychoendocrine research on the pituitary-adrenal cortical system. Psychosom Med. 1968 Sep-Oct;30(5):Suppl:576-607. No abstract available. PMID 4303377
- [Background] Weiss JM. Somatic effects of predictable and unpredictable shock. Psychosom Med. 1970 Jul-Aug;32(4):397-408. doi: 10.1097/00006842-197007000-00008. No abstract available. PMID 5535207
- [Background] Pawlak CR, Jacobs R, Mikeska E, Ochsmann S, Lombardi MS, Kavelaars A, Heijnen CJ, Schmidt RE, Schedlowski M. Patients with systemic lupus erythematosus differ from healthy controls in their immunological response to acute psychological stress. Brain Behav Immun. 1999 Dec;13(4):287-302. doi: 10.1006/brbi.1999.0553. PMID 10600217
- [Background] Schedlowski M, Hosch W, Oberbeck R, Benschop RJ, Jacobs R, Raab HR, Schmidt RE. Catecholamines modulate human NK cell circulation and function via spleen-independent beta 2-adrenergic mechanisms. J Immunol. 1996 Jan 1;156(1):93-9. PMID 8598500
- [Background] Schmid-Ott G, Jacobs R, Jager B, Klages S, Wolf J, Werfel T, Kapp A, Schurmeyer T, Lamprecht F, Schmidt RE, Schedlowski M. Stress-induced endocrine and immunological changes in psoriasis patients and healthy controls. A preliminary study. Psychother Psychosom. 1998;67(1):37-42. doi: 10.1159/000012257. PMID 9491439
- [Derived] Doering BK, Wegner A, Hadamitzky M, Engler H, Rief W, Schedlowski M. Effects of Neurexan (R) in an experimental acute stress setting--An explorative double-blind study in healthy volunteers. Life Sci. 2016 Feb 1;146:139-47. doi: 10.1016/j.lfs.2015.12.058. Epub 2016 Jan 7. PMID 26772822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out in 2 outpatient clinics in Germany (Marburg and Essen).
Pre-assignment Details: All 66 healthy participants were enrolled and none of them was excluded prior to randomization.
Groups:
- Neurexan®: 0.6 mg / tablet, 6 tablets, 1 tablet every 30 minutes from -180 minutes to -30 minutes
  Neurexan®
- Placebo: 6 tablets, 1 tablet every 30 minutes from -180 minutes to -30 minutes
  Placebo
Period: Overall Study
Arm/Group | Neurexan® | Placebo
Started | 34 | 32
Completed | 34 | 30
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. Two premature terminators could not be evaluated for primary efficacy, so 34 participants in the Neurexan group and 30 participants in the Placebo group formed the Full Analysis Set for analysis of efficacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurexan® | Placebo | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (7.0) | 40.7 (8.2) | 40.9 (7.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 66
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants] — 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. Two premature terminators could not be evaluated for primary efficacy, so 34 participants in the Neurexan group and 30 participants in the Placebo group formed the Full Analysis Set for analysis of efficacy.
  participants
    Germany | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Acute Stress Measured by Tension
Description: Tension and nervousness were self-assessed by the participants on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) before and after a stress test. The VAS is used to determine the subjective impression of tension and nervousness on a 10 cm bipolar visual scale ranging from 0
  = "not at all" to 100 = "highly". The measurements started with first intake of Neurexan or Placebo and were repeated until 100 minutes after the end of the stress test. The total stress was then summarized with the area under the curve (AUC) method.
Time Frame: -210 minutes to +100 minutes
Population: 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. 34 Neurexan and 30 Placebo participants that could be evaluated for primary efficacy formed the Full Analysis Set for analysis of efficacy.
Measure: Median (Full Range); unit: mm*min
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
mm*min | 3335.7 [345 to 16411] | 3360.3 [0 to 21115]
Statistical Analysis 1: Comparison: Neurexan® vs Placebo; The null-hypotheses of no treatment differences were tested by the two-sided t-tests from the respective ANCOVAs; Test type: Superiority or Other; p = 0.7726, ANCOVA — Threshold less than or equal to 0.05. The final analysis demonstrated reasonable doubt of the implicit normality assumption of the two sets of AUC data, thus medians presented for efficacy analysis. Need for further investigation (ex-post analyses)

2. Primary Outcome: Acute Stress Measured by Nervousness
Description: as for outcome 1
Time Frame: -210 minutes to +100 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: mm*min
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
mm*min | 3147.4 [247 to 17050] | 3022.5 [0 to 21409]
Statistical Analysis 1: Comparison: Neurexan® vs Placebo; The null-hypotheses of no treatment differences were tested by the two-sided t-tests from the respective ANCOV As; Test type: Superiority or Other; p = 0.5702, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Changes in Saliva Alpha Amylase
Description: The stress biomarkers plasma and saliva cortisol, alpha amylase, Adrenocorticotropic Hormone and catecholamines (norepinephrine and epinephrine) were measured before and after a stress test. The measurements started 60 minutes before stress test and were repeated until 100 minutes after the end of the stress test.
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: IU/mL
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
IU/mL
  - 60 min | 112.9 [19.7 to 353.7] | 133.3 [23.7 to 421.1]
  +15 min | 201.9 [78.4 to 729.7] | 216.0 [49.3 to 670.9]
  +45 min | 140.8 [25.6 to 420.4] | 142.1 [37.1 to 484.8]
  +100 min | 149.9 [29.2 to 465.1] | 140.6 [35.1 to 417.3]

4. Secondary Outcome: Changes in Saliva Cortisol
Description: The stress biomarkers plasma and saliva cortisol and alpha amylase and Adrenocorticotropic Hormone and catecholamines (norepinephrine and epinephrine) were measured before and after a stress test. The measurements started 60 minutes before stress test and were repeated until 100 minutes after the end of the stress test.
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: nmol/mL
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
nmol/mL
  - 60 min | 7.1 [3.0 to 17.4] | 7.1 [2.7 to 32.4]
  +15 min | 19.4 [7.2 to 120.8] | 20.0 [6.1 to 86.6]
  +45 min | 15.3 [7.0 to 80.7] | 21.2 [3.9 to 81.4]
  +100 min | 6.4 [3.7 to 20.9] | 8.9 [3.6 to 21.2]

5. Secondary Outcome: Changes in Plasma Adrenocorticotropic Hormone (ACTH)
Description: as for outcome 4
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. For evaluation of plasma ACTH, 31 Neurexan and 29 Placebo participants were evaluated due to insufficient sample.
Measure: Median (Full Range); unit: ng/L
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 31 | 29
ng/L
  - 60 min | 22.5 [9.2 to 330.4] | 19.1 [5.5 to 493.2]
  +15 min | 37.7 [13.9 to 124.2] | 37.0 [13.6 to 209.7]
  +45 min | 20.3 [7.5 to 42.3] | 20.7 [7.5 to 79.4]
  +100 min | 11.3 [3.2 to 24.4] | 10.7 [5.4 to 24.0]

6. Secondary Outcome: Changes in Plasma Cortisol
Description: as for outcome 4
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. For evaluation of plasma Cortisol, 31 Neurexan and 29 Placebo participants were evaluated due to insufficient sample.
Measure: Median (Full Range); unit: nmol/L
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 31 | 29
nmol/L
  - 60 min | 331.6 [97.6 to 614.8] | 325.5 [54.2 to 1006.7]
  +15 min | 441.1 [281.4 to 987.1] | 569.8 [174.1 to 1048.7]
  +45 min | 403.1 [223.7 to 1260] | 535.4 [142.5 to 841.2]
  +100 min | 228.4 [94.6 to 671.8] | 273.3 [108.5 to 658.0]

7. Secondary Outcome: Changes in Plasma Catecholamines (Epinephrine)
Description: as for outcome 4
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. For evaluation of plasma Epinephrine, 30 Neurexan and 26 Placebo participants were evaluated due to insufficient sample.
Measure: Median (Full Range); unit: ng/L
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 30 | 26
ng/L
  - 60 min | 42.6 [10.0 to 98.0] | 35.6 [8.1 to 146.0]
  +15 min | 32.9 [10.0 to 116.0] | 47.4 [10.0 to 126.0]
  +45 min | 41.4 [10.0 to 152.0] | 26.4 [10.0 to 101.0]
  +100 min | 31.9 [0.0 to 91.3] | 41.1 [11.3 to 89.9]

8. Secondary Outcome: Changes in Plasma Catecholamines (Norepinephrine)
Description: as for outcome 4
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: 34 participants were randomized to Neurexan and 32 participants to Placebo and all randomized participants were included in the Safety Set. For evaluation of plasma Norepinephrine, 30 Neurexan and 26 Placebo participants were evaluated due to insufficient sample.
Measure: Median (Full Range); unit: ng/L
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 30 | 26
ng/L
  - 60 min | 463.0 [99 to 990] | 457.0 [253 to 1329]
  +15 min | 584.0 [150 to 1352] | 591.5 [316 to 1856]
  +45 min | 481.0 [231 to 1530] | 476.0 [168 to 1189]
  +100 min | 451.5 [215 to 1318] | 482.5 [230 to 815]

9. Secondary Outcome: Changes in Natural Killer (NK) Cells (Subgroup)
Description: The Natural Killer Cells as immune cells and stress biomarkers were measured before and after a stress test. The measurements started 60 minutes before stress test and were repeated until 100 minutes after the end of the stress test.
Time Frame: -60 minutes, +15 minutes, +45 minutes, +100 minutes
Population: The test was only conducted in the Essen site where 15 participants randomized to Neurexan and 16 participants randomized to Placebo could be evaluated for NK cells.
Measure: Median (Full Range); unit: percentage of lymphocytes
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 15 | 16
percentage of lymphocytes
  - 60 min | 13.5 [5.5 to 23.2] | 11.65 [6.3 to 21.0]
  +15 min | 21.00 [9.1 to 36.2] | 20.40 [8.0 to 37.3]
  +45 min | 10.30 [3.3 to 20.4] | 9.10 [5.4 to 18.6]
  +100 min | 13.10 [4.3 to 20.9] | 8.65 [5.5 to 21.5]

10. Secondary Outcome: Changes in Blood Pressure
Description: Blood pressure and heart rate were measured before and after a stress test by continuous cardiovascular recording.
  The measurements started 30 minutes before stress test and were repeated until 45 minutes after the end of the stress test.
Time Frame: -15 minutes, 0 minutes, +15 minutes, +45 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
mmHg
  Systolic -15 min | 122.0 [96 to 153] | 123.5 [102 to 147]
  Systolic 0 min | 132.0 [106 to 201] | 142.0 [110 to 168]
  Systolic +15 min | 125.0 [99 to 164] | 133.5 [105 to 153]
  Systolic +45 min | 121.5 [96 to 163] | 125.0 [101 to 182]
  Diastolic - 15 min | 79.5 [58 to 109] | 81.5 [61 to 98]
  Diastolic 0 min | 81.0 [66 to 117] | 91.0 [63 to 107]
  Diastolic +15 min | 83.5 [65 to 115] | 89.0 [63 to 109]
  Diastolic +45 min | 81.0 [34 to 113] | 83.0 [63 to 113]

11. Secondary Outcome: Changes in Heart Rate
Description: as for outcome 10
Time Frame: -15 minutes, 0 minutes, +15 minutes, +45 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: beats per minute
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
beats per minute
  -15 min | 70.0 [55 to 96] | 69.0 [52 to 94]
  0 min | 88.0 [65 to 115] | 89.5 [65 to 131]
  +15 min | 69.5 [56 to 94] | 71.0 [53 to 119]
  +45 min | 71.0 [59 to 106] | 71.0 [55 to 91]

12. Secondary Outcome: State Anxiety and Stress Perception Measured by STAI-X1
Description: State anxiety and stress perception were measured by State-Trait Anxiety Inventory X1 before and after a stress test. The measurements took place 90 minutes before the stress test and were repeated at 15 and 100 minutes after the end of the stress test. The German version of the State-Trait-Anxiety Inventory was used and differentiates between temporary/emotional state anxiety versus personality trait anxiety. The two scales with 20 items each assess (1) anxiety as a trait (STAI-X2) and (2) anxiety as a state (STAI-XI). Answers are given in a 4-point rating scale ranging from 1 ="not at all" to 4 ="very true". For analysis of each, STAI-scale single scores were summed up to one total score, representing the state and trait anxiety. Score range is 20-80 and higher scores indicate a higher anxiety.
Time Frame: -90 minutes, +15 minutes, +100 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
units on a scale
  - 90 min | 31.0 [21 to 45] | 29.5 [22 to 50]
  +15 min | 54.5 [24 to 74] | 51.5 [23 to 68]
  +100 min | 33.0 [20 to 69] | 31.5 [22 to 48]

13. Secondary Outcome: Psychological Questionnaire (Modified Somatic SCL90)
Description: The SCL90 has 90 items with dimensions like depression, somatization, obsessive-compulsive disorder, social insecurity, anxiety, phobic anxiety, aggression/hostility, paranoid ideation, psychoticism and each item in a subscale ranged from 0 to 4. The lower range values are favorable outcomes and higher are worse outcomes. The modified somatic SCL90 uses the SCL90 somatization items, but instead of a 7 day timeframe asks for "now". The corresponding items from SCL90 were: 1, 4, 12, 27, 40, 42, 48, 49, 52, 53, 56, 58 and the introductory question: "How much do you currently suffer from" ("Wie sehr leiden Sie momentan unter:"). The median of the average Modified Somatic SCL90 score is reported. The average score was calculated at each time point as the sum score divided by the number of non-missing individual question results for subjects with no more than 2 missing responses. The lower values in the range represent favorable outcomes while the higher values represent worse outcomes.
Time Frame: -210 minutes, +100 minutes
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Neurexan® | Placebo
Number analyzed (Participants) | 34 | 30
units on a scale
  - 210 min | 0.000 [0.00 to 0.83] | 0.000 [0.00 to 0.42]
  +100 min | 0.000 [0.00 to 0.75] | 0.000 [0.00 to 0.33]

ADVERSE EVENTS:
Time Frame: Randomization until individual study end
Description: All adverse events that occurred after the participant has received at least one dose of the product under investigation were to be collected and reported
Arm/Group | Neurexan® | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 4/34 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neurexan® (N=34) | Placebo (N=32)
Tremor (Nervous system disorders) | 0 | 1
Feeling Cold (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Procedural dizziness (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Blood Pressure Decrease (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agreements are in place restricting the PI from independently publishing the study results. Currently working with both PIs on several publications of the NEUPRO studies.